CLINICAL TRIAL: NCT06654310
Title: The Fundamentals of Communication in Surgery (FCS): A Pilot Study to Evaluate the Scalability and Impact of A Clinical Communication Curriculum
Brief Title: The Fundamentals of Communication in Surgery
Acronym: FCS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Josiah Macy, Jr. Foundation (Unknown); University of Oklahoma (Other); University of Pittsburgh (Other); University of South Florida (Other); West Virginia University (Other); Duke University (Other); Association for Academic Surgery (Unknown); Inova Fairfax Medical Campus (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-0620; A539750 (Other: UW- Madison)
Record Dates: First submitted 2024-10-09; First posted 2024-10-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Communication Research; Communication Programs
Keywords: Surgical Trainees; Fundamentals of Communication in Surgery; FCS; Best Case/Worst Case; BC/WC; Better Conversations
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Learners: All general surgery trainees at each institution will have access to the training program as part of their regularly scheduled educational curriculum, regardless of training year or status as a categorical resident.
  Interventions: Behavioral: Delivery of FCS Skills Curriculum

INTERVENTIONS:
Behavioral: Delivery of FCS Skills Curriculum — The UW study team will conduct two 2-hour train-the-trainer sessions with all surgical attendings who have committed to participation as a trainer in the FCS curriculum. The designated trainer will deliver each 2-hour session during the existing formal educational time for residents. If existing protected educational time will not allow for a 2-hour training session, the sessions can be delivered in two 1-hour sessions. These sessions will be incorporated into the curriculum similar to all other formal training provided to residents with the same expectations to attend.
  Each 2-hour FCS session starts with a 30-minute exercise in empathic communication. The remaining 90 minutes are devoted to skills that support decision making about surgery.

SUMMARY:
The goal of this observational study is to evaluate the impact of the FCS curriculum on achieving the learning objectives and resident reported self-efficacy with communication skills and determine the scalability of the training across a range of general surgery training programs

DETAILED DESCRIPTION:
The researchers have developed a 5-year curriculum for surgical trainees called the Fundamentals of Communication in Surgery (FCS). The training includes core communication skills, e.g., expressing empathy, and frameworks to support informed consent and serious illness conversations, specifically Best Case/Worst Case and Better Conversations. The curriculum provides one developmentally appropriate two-hour session for each of the five years of surgical training. Because the training is skills based (e.g., scenario planning) and not procedure based (e.g., goals of care conversations) exercises are focused on specific techniques that build over subsequent sessions.

Researchers will invite 1-3 surgical attendings per site with an interest in surgical education to serve as trainers for the FCS curriculum.

All general surgery trainees at each institution will have access to the training program as part of their regularly scheduled educational curriculum, regardless of training year or status as a categorical resident. If there is interest, researchers will provide access to the curriculum to fellows and residents in affiliated programs, e.g., plastic surgery.

Researchers will invite site personnel who have roles related to surgical education including the program director and associate program director (if applicable), 2 to 3 attending surgeons who have high contact with residents in urgent care settings (e.g., emergency general surgery), 1 to 2 members of the education coordination team.

ELIGIBILITY:
Inclusion Criteria:

* surgical attendings with an interest in surgical education
* surgery trainees

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be from each participating site.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Trainee Reaction to the Training | Day of training through 2 months post-training
  Surgical trainees will complete a 5-item survey on a scale of 1-5 (1= strongly disagree, 5= strongly agree). Total scores range from 5-25, with higher scores indicating greater acceptability of the curriculum.

SECONDARY OUTCOMES:
Trainee Self-Efficacy - Ability | Before training, directly after training, and 2 months post-training
  Surgical trainees will complete an 8-item ability survey on a scale of 1-5 (1= not at all able to do, 5= easily able to do). Total scores range from 8-40, with higher scores indicating a better ability to communicate.
Receipt of Curriculum | 1 day of training
  Educational coordinators will provide a direct count of the number of categorical residents who attend their session, divided by the total number eligible to attend.
Performance of Skills | Baseline (before training), directly after training, and 2 months post-training
  Trainers will observe surgical trainees to evaluate them on various items using a scoring rubric. Each item will be scored as not done, done, or exceptional.
  Binary Scoring (0/1) 0: Not Done
  1: Done
  Ternary Scoring (0/1/2) 0: Not Done
  1. Done
  2. Exceptional
Fidelity to the Intervention | 1 day of training
  A member of the UW study team will travel to each institution once to observe one 2-hour educational session in person. The observer will use an implementation checklist (rubric) to record performance of discrete elements of the curriculum and the fidelity to the overall training program goals as described in the learning objectives.
Trainee Self-Efficacy - Preparedness | Before training, directly after training, and 2 months post-training
  Surgical trainees will also complete a 6-item preparedness survey with a scale of 1-5 (1= not at all prepared, 5= very well prepared). Total scores range from 6-35, with higher scores indicating greater confidence in navigating treatment decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret (Gretchen) L Schwarze, MD, MPP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No